CLINICAL TRIAL: NCT00792467
Title: Phase II Trial of the Histone-Deacetylase Inhibitor ITF2357 Followed by Mechlorethamine in Relapsed/Refractory Hodgkin's Lymphoma Patients
Brief Title: Trial of the Histone-Deacetylase Inhibitor ITF2357 Followed by Mechlorethamine in Relapsed/Refractory Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Italfarmaco (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DSC/07/2357/31; 2007-007091-41 (EudraCT Number)
Record Dates: First submitted 2008-11-17; First posted 2008-11-18 (Estimated); Results first posted 2021-04-19 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-04

CONDITIONS: Hodgkin's Lymphoma
MeSH Terms: conditions — Hodgkin Disease | interventions — givinostat hydrochloride; givinostat; Histone Deacetylase Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ITF2357 (Experimental): Patients received the following therapy cycle
  * ITF2357, 50 mg every 6 hours, per os, days 1 - 3;
  * Mechlorethamine, 6 mg/sqm, intravenously , day 4. Therapy was administered every 21 days as long as there was no evidence of progressive disease or unacceptable toxicity, but in any case for a maximum of 12 cycles.
  The mean number of complete treatment cycles received by patients was 5.25, with a minimum of 1 cycle and a maximum of 12 cycles.
  Interventions: Drug: ITF2357

INTERVENTIONS:
Drug: ITF2357 — ITF2357, supplied as hard gelatine capsules for oral administration at the strength of 50 mg each.
  Other Names: Givinostat, histone deacetylase inhibitor

SUMMARY:
This study has the following objectives:

Primary Objective

* To evaluate the anti-lymphoma efficacy of daily oral doses of ITF2357 followed by intravenous Mechlorethamine administered to patients with refractory/relapsed Hodgkin's lymphoma.

Secondary Objective

- To evaluate the safety and tolerability of multiple courses of ITF2357 followed by Mechlorethamine in a population of chemotherapy pretreated patients.

DETAILED DESCRIPTION:
This is a single-center, open label, phase II study aimed at testing the activity of multiple cycles of ITF2357 followed by Mechlorethamine administered to patients with relapsed/refractory Hodgkin's lymphoma.

Patients will receive a maximum of twelve 3-week cycles of ITF2357 followed by Mechlorethamine according to the following schema:

* ITF2357, 50 mg every 6 hours, per os, days 1 - 3
* Mechlorethamine, 6 mg/sqm, intravenously , day 4 Study therapy will be administered every 21 days as long as there is no evidence of progressive disease or unacceptable adverse events or patient's request to discontinue treatment occurs, but in any case for a maximum of 12 cycles.

Decision regarding the continuation of ITF2357/Mechlorethamine therapy will be made on (i)the basis of tumor reassessment following cycles 2, 6, 9, and 12 and (ii) the occurrence of toxicity. Tumor response will be evaluated according to the International Working Group response criteria HL.

Treatment will be administrated on an outpatient basis and patients will be followed regularly with physical and laboratory tests, as specified in the protocol; in case of hospitalisation, the treatment will be continued or interrupted according to the Investigators' decision.

The study will accrue 23 patients evaluable for efficacy and the anticipated duration of the study is about 24 months.

Histone deacetylases (HDACs) are enzymes involved in the remodeling of chromatin, and have a key role in the epigenetic regulation of gene expression. In addition, the activity of non-histone proteins can be regulated through HDAC-mediated hypoacetylation. In recent years, inhibition of HDACs has emerged as a potential strategy to reverse aberrant epigenetic changes associated with cancer, and several classes of HDAC inhibitors have been found to have potent and specific anticancer activities in preclinical studies.

Hodgkin's lymphoma (HL) is a relatively uncommon lymphoma histotype, with an incidence in Italy of approximately 1700 new cases per year (approximately 12% of all lymphomas). Combination chemotherapy with or without radiotherapy cures approximately 70 percent of advanced-stage HL. Fifty percent of the failing patients can be salvaged by second line chemotherapy (mainly high-dose regimens), while the remaining patients eventually die by disease progression. The development of an effective salvage regimen for this refractory/resistant population represents a true unmet medical need.

The use in the latter patient subset of HDAC inhibitors, like ITF2357, is supported by several considerations. Namely: (1) a related hydroxamate, SAHA, has shown activity in this clinical condition; (2) the drug markedly inhibits the production of several cytokines, and cytokine production in HL granuloma has a defined role in the pathogenesis of HL; (3) an effective treatment for refractory/relapsed HL is presently lacking; (4) ITF2357, up to 200 mg daily per os, has shown a favorable toxicity profile. All the above mentioned arguments represent a strong rationale prompting the use of ITF2357 in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Written Informed Consent;
* Age ≥18 years;
* Histologically confirmed diagnosis of Hodgkin's lymphoma;
* Subjects who have failed second-line or subsequent-line salvage chemo- radiotherapy regimens for whom no other treatment options of proven efficacy can be given;
* Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements;
* ANC ≥1500/µL; Platelet count ≥75000/µL;
* Hemoglobin ≥9 g/dL (may not be transfused or treated with erythropoietin to maintain or exceed this level);
* Total bilirubin ≤1.6 mg/dL; AST or ALT ≤2.5 times the upper limit of normal;
* Serum creatinine ≤2.0 mg/dL or creatinine clearance >50 mL/min;
* Serum Potassium and Magnesium within normal limits;
* Subjects with at least one bi-dimensional lesion measurable by CT-scan or MRI, according to the Revised Response Criteria for Malignant Lymphoma of the International Working Group (J Clin Oncol, 25:579-586, 2007);
* ECOG performance status of 0 or 1;
* Use of an effective means of contraception for women of childbearing potential and men with partners of childbearing potential;
* Life expectancy of >3 months;
* Subjects receiving intravenous Mechlorethamine (6 mg/sqm) as single agent at least 4 weeks before study entry;
* Willingness and capability to comply with the requirements of the study.

Exclusion Criteria:

* Active bacterial or mycotic infection requiring antimicrobial treatment
* Pregnancy or lactation
* Anticancer chemotherapy or radiotherapy during the study or within 4 weeks of study entry.
* A marked baseline prolongation of QT/QTc interval (e.g. repeated demonstration of a QTc interval > 450 ms, according to Bazett's correction formula - see appendix I for the formula)
* Use of concomitant medications that prolong the QT/QTc interval (see appendix H for full list)
* Clinically significant cardiovascular disease including:
* Uncontrolled hypertension, myocardial infarction, unstable angina
* New York Heart Association (NYHA) Grade II or greater congestive heart failure
* History of any cardiac arrhythmia requiring medication (irrespective of its severity)
* A history of additional risk factors for TdP (e.g., heart failure, hypokalemia, family history of Long QT Syndrome)
* Positive blood test for HIV, HBV and HCV
* Identification of viral DNA by quantitative PCR for EBV and JC virus.
* History of other diseases, metabolic dysfunctions, physical examination findings, or clinical laboratory findings giving reasonable suspicion of a disease or condition that contraindicates use of an investigational drug or that might affect interpretation of the results of the study or render the subject at high risk from treatment complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-02; Primary Completion 2010-07 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Massimo Gianni, MD, Principal Investigator — Istituto Nazionale per la Cura e lo Studio dei Tumori, Milano, Italy
Locations (1):
- Istituto Nazionale per la Cura e lo Studio dei Tumori, Milan, Italy

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients enrolled were 24 subjects of both genders, age ≥18 years, with histologically confirmed diagnosis of Hodgkin's lymphoma and refractory or relapsed.
Groups:
- ITF2357: Patients received the following therapy cycle
  * ITF2357, 50 mg every 6 hours, per os, days 1 - 3;
  * Mechlorethamine, 6 mg/sqm, intravenously , day 4. Therapy was administered every 21 days as long as there is no evidence of progressive disease or unacceptable toxicity, but in any case for a maximum of 12 cycles.
  ITF2357: ITF2357, supplied as hard gelatine capsules for oral administration at the strength of 50 mg each.
Period: Overall Study
Arm/Group | ITF2357
Started | 24
Completed | 2
Not Completed | 22
Not completed — progression of disease | 17
Not completed — Adverse Event | 1
Not completed — patient request | 1
Not completed — Lost to Follow-up | 1
Not completed — Patient achieved a PR and allogenic transplant was performed | 1
Not completed — Patient in CR and HLA-matched donor available. Allogenic SCT performed | 1

BASELINE CHARACTERISTICS:
Groups:
- ITF2357: Patients will receive the following therapy cycle
  * ITF2357, 50 mg every 6 hours, per os, days 1 - 3;
  * Mechlorethamine, 6 mg/sqm, intravenously , day 4. Therapy will be administered every 21 days as long as there is no evidence of progressive disease or unacceptable toxicity, but in any case for a maximum of 12 cycles.
  ITF2357: ITF2357, supplied as hard gelatine capsules for oral administration at the strength of 50 mg each.
Arm/Group | ITF2357
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.83 (14.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Italy | 24

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: OR rate among patients treated is defined according to the Revised Response Criteria for Malignant Lymphoma of the International Working Group.
  In medicine, a response rate is the percentage of patients whose cancer shrinks or disappears after treatment.
  The FDA definition of ORR is the proportion of patients with tumor size reduction of a predefined amount and for a minimum time period.
  The tumor objective response rate (ORR) is an important parameter to demonstrate the efficacy of a treatment in oncology.
  The ORR is valuable for clinical decision making in routine practice and a significant end-point for reporting the results of clinical trials.
Time Frame: At each 21-day cycle for a maximum of 12 cycles
Population: Intent-to-treat population: all patients valid for Safety population. Per Protocol population: all recruited patients who: 1) were not severe protocol violators; 2) had at least one on-study tumor assessment beside baseline; 3) experienced disease progression or, if not, received at least 2 cycles of the study treatment consecutively.
Measure: Number; unit: percentage of patients
Groups:
- ITT Population; PP Population: Patients received the following therapy cycle
  * ITF2357, 50 mg every 6 hours, per os, days 1 - 3;
  * Mechlorethamine, 6 mg/sqm, intravenously , day 4. Therapy was administered every 21 days as long as there is no evidence of progressive disease or unacceptable toxicity, but in any case for a maximum of 12 cycles.
  ITF2357: ITF2357, supplied as hard gelatine capsules for oral administration at the strength of 50 mg each.
Arm/Group | ITT Population | PP Population
Number analyzed (Participants) | 24 | 16
percentage of patients
  Objective Response achieved | 25.00 | 37.50
  Objective Response not achieved | 75.00 | 62.50

2. Primary Outcome: Proportion of Responders (Complete -CR- or Partial PR-)
Description: Complete responder (CR) and partial responder (PR) among patients treated are defined according to the Revised Response Criteria for Malignant Lymphoma of the International Working Group.
  CR is defined as complete disappearance of all detectable clinical evidence of disease and disease-related symptoms if present before therapy.
  PR is defined as regression of measurable disease and no new sites. The frequencies of patients achieving objective response (i.e. subjects whose best overall response was CR or PR) and the frequencies of patients who did not achieve an objective response (i.e.subjects whose best overall response was equal to stable disease - SD, progressive disease - PD - or not evaluable) in ITT and PP populations are reported.
  NED= no evidence of disease
Time Frame: At each 21-day cycle for a maximum of 12 cycles
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | ITT Population | PP Population
Number analyzed (Participants) | 24 | 16
percentage of participants
  CR/NED | 4.17 | 6.25
  PR | 20.83 | 31.25
  SD | 29.17 | 25.00
  PD | 37.50 | 37.50
  Not evaluable | 8.33 | 0

3. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS is defined as the time from the 1st day of the 1st cycle of treatment until objective tumor progression or death. It included deaths, thus could be correlated to overall survival. If a patient did not have disease progression, PFS was censored at the date of last available tumor assessment (including those at end of study or follow-up visit).
Time Frame: From the first day of the first cycle of treatment until objective tumor progression or death, whichever came first, assessed up to 450 days from the start of the first cycle of treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | ITT Population | PP Population
Number analyzed (Participants) | 24 | 16
Days | 164.53 (28.66) | 183.94 (39.38)

4. Secondary Outcome: Time To Response (TTR)
Description: TTR is defined as the time from the 1st day of the 1st cycle until the date of achieving a response (CR or PR).
  In case of no objective response, TTR was censored at the date of last available tumor assessment (including those at end of study or follow-up visit).
Time Frame: From the first day of the first cycle until the date of achieving a response assessed up to 250 days from the start of the first cycle of treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | ITT Population | PP Population
Number analyzed (Participants) | 24 | 16
Days | 123.52 (11.70) | 114.34 (14.81)

5. Secondary Outcome: Response Duration (RD):
Description: Duration of objective response (CR or PR) was applied only to patients whose best overall response was CR or PR.
Time Frame: From the first day of the first cycle of treatment until objective tumor progression or death, whichever came first, or last available tumor assessment (assessed up to 350 days from the start of the first cycle of treatment).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | ITT Population | PP Population
Number analyzed (Participants) | 6 | 6
Days | 199.96 (42.77) | 199.96 (42.77)

ADVERSE EVENTS:
Time Frame: Throughout the course of the study, up to a maximum of 12 cycles, an average of 1 year.
Arm/Group | ITF2357
All-Cause Mortality (participants affected / at risk) | 3/24
Serious Adverse Events (participants affected / at risk) | 1/24
Other Adverse Events (participants affected / at risk) | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ITF2357 (N=24)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fever (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ITF2357 (N=24)
Anaemia (Blood and lymphatic system disorders) | 12
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Leukopenia (Cardiac disorders) | 1
Neutropenia (Cardiac disorders) | 11
Thrombocytopenia (Cardiac disorders) | 16
Atrial fibrillation (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 5
Dysphagia (Gastrointestinal disorders) | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 7
Stomatitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 5
Asthenia (General disorders) | 6
chest pain (General disorders) | 1
Extravasation (General disorders) | 1
Fatigue (General disorders) | 1
Injection site reaction (General disorders) | 1
Pyrexia (General disorders) | 7
Graft versus host disease (Immune system disorders) | 1
Infection (Infections and infestations) | 2
Skin infection (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 3
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3
Butterfly rash (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 2
Deep vein thrombosis (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No